CLINICAL TRIAL: NCT06445803
Title: A Preliminary Study to Evaluate the Safety, Tolerability, Preliminary Efficacy and Pharmacokinetic Profile of KQ-2002 (CD19/CD22 CAR-T) in Adults With Recurrent or Refractory Acute Lymphoblastic Leukemia or Non-Hodgkin's Lymphoma
Brief Title: CD19/CD22 CAR-T Cells in Adults With R/R ALL or NHL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rong Tao (Other)
Collaborators: Novatim Immune Therapeutics (Zhejiang) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Rong Tao, Chief physician, Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQ-2002-XC001
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia With Failed Remission; B-cell Lymphoma Refractory; B-cell Lymphoma Recurrent
Keywords: CAR-T therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): CD19/CD22-CAR-transduced T cells at escalating doses (0.5~5.0 ×10^6 cells/kg)
  Interventions: Biological: KQ-2002 CAR-T cells （CD19/CD22 CAR T-Cells）
- Dose expansion (Experimental): CD19/CD22-CAR-transduced T cells at MTD or highest dose administered
  Interventions: Biological: KQ-2002 CAR-T cells （CD19/CD22 CAR T-Cells）

INTERVENTIONS:
Biological: KQ-2002 CAR-T cells （CD19/CD22 CAR T-Cells） — CD19/CD22 cells will be infused on Day1 after induction chemotherapy regimen.
  Lymphodepleting chemotherapy:3 days of IV chemotherapy with fludarabine and cyclophosphamide.
  Fludarabine 30 mg/m2/day IV x 4 days (days -5 through -3) Cyclophosphamide 500 mg/m2/day IV x 2 days (days -5 and-3)

SUMMARY:
This study examines the safety, tolerability and preliminary efficacy of anti-CD19 /CD22 CAR T cells (KQ-2002)manufactured on-site in adults with relapsed or refractory CD19+ B cell acute lymphoblastic leukemia or CD19+ B cell non Hodgkin lymphoma.

DETAILED DESCRIPTION:
Patients will undergo screening, leukapheresis (cell collection), lymphodepleting chemotherapy with fludarabine and cyclophosphamide, followed by the anti-CD19 KQ-2002 CAR T cell infusion. The lymphodepleting chemotherapy is administered over 3 days IV to prepare the body for the CAR T cells. The CAR-T cells are infused between 2-7 days after the last dose of chemotherapy. Patients will be followed for two years after the cell infusion on the study and for up to 15 years to monitor for potential long term side effects of cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,≥18 years old;
* Histologically confirmed diagnosis of B-ALL or B-NHL(meeting one of the following conditions):

(B-NHL)

1. Second or greater relapse (CD20 regimens must be included) OR
2. Refractory to first-line chemotherapy or relapse within 1 year OR
3. Relapse within 1 year of auto-HSCT.
4. With measurable or evaluable lesions（Dose expansion cohort） (B-ALL)

a. Relapse within 12 months of complete remission on first treatment OR b. Relapse after second-line treatment OR c. Relapse after auto HST OR d. Failure to achieve CR/CRi at the end of induction therapy OR e. Ph+ ALL intolerance to TKI or refractory or relapse after treatment with at least two and more TKIs.

* ECOG 0~2
* Estimated survival time ≥ 12 weeks;
* Main tissues and organs function well.

Exclusion Criteria:

* Subjects will be excluded related to the following prior therapy criteria:Prior treatment with bendamustine-containing or fludarabine;Anti-T-cell monoclonal antibody, donor lymphocyte infusion, and CNS radiotherapy within 8 weeks; Chemotherapy, lenalidomide, bortezomib within 2 weeks; vincristine within 1 week; glucocorticoids (prednisone ≥7.5 mg/d or equivalent) within 72 h
* Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening), or any uncontrolled infection at screening
* Uncontrolled, symptomatic, intercurrent illness including but not limited to angina pectoris, cerebrovascular accident or transient ischemia (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), New York Heart Association (NYHA) classification of ≥ Class III congestive heart failure, severe arrhythmia poorly controlled by medications, hepatic, renal, or metabolic disorders, and hypertension that is uncontrolled by standard therapy；
* active bleeding, or venous thromboembolic event
* Autoimmune diseases (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, etc.) that result in end-organ damage or require systemic application of immunosuppressive drugs
* Central nervous system (CNS) disease or symptoms of CNS involvement
* Pregnant or nursing (lactating) women
* Presence of Grade 2 or above non-hematologic toxicity , alopecia and grade 2 neuropathy excluded
* Any Iinappropriate conditions in the opinion of the PI .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-limiting toxicity | Up to 28 days
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Incidence and severity of adverse events | Up to 15 years
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Overall response rate | up to 15 years
  Proportion of patients achieving a response
Progression free survival | up to 15 years
  Preparative regimen until the documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival | up to 15 years
  Overall survival (OS) will be determined as the time from the start of the preparative regimen until death
MRD negative response rates（ Acute Lymphoblastic Leukemia ） | up to 15 years
  MRD status post infusion，MRD will be performed utilizing flow cytometry or PCR.
Persistence of CD19/CD22 CAR-T cells blood, bone marrow | up to 15 years
  pk properties of CD19/CD22 CAR-T

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanchang University;, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No